CLINICAL TRIAL: NCT02420275
Title: Controlled Randomized Trial Estimating the Efficiency of Blue Enriched White Light on Sequel Fatigue, in Victims of Severe Cranial Traumas
Brief Title: Trial Estimating the Efficiency of the Light Therapy in Brain Trauma Sequel Fatigue
Acronym: phototrauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Garches (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A000321-48
Record Dates: First submitted 2015-04-10; First posted 2015-04-17 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-02

CONDITIONS: Diffuse Brain Injury
Keywords: brain injury; blue enriched withe bright light therapy; sequel fatigue
MeSH Terms: conditions — Brain Injuries, Diffuse; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Severe brain injury patient (Placebo Comparator): Severe brain injury patients with placebo
  Interventions: Other: placebo
- Severe brain injury patient with device (Experimental): Severe brain injury patients withe with "Luminette",Lucimed Belgium
  Interventions: Device: "Luminette",Lucimed Belgium

INTERVENTIONS:
Other: placebo — THIS GROUP WILL RECEIVE NO BRIGHT LIGHT
  Arms: Severe brain injury patient
Device: "Luminette",Lucimed Belgium — THIS GROUP WILL RECEIVE BLEU LIGHT ENRICHIDED IN WITHE BRIGHT LIGHT
  Arms: Severe brain injury patient with device

SUMMARY:
After a brain injury (BI) , patients complain in particular about sequel fatigue. This symptom affects about 50 % of the patients; it is severe, with a repercussion on quality of life, reeducation and occupational reintegration, and persists often at a distance of the accident. The investigators' hypothesis is that patients who presented a severe BI could benefit from a treatment by withe blue enriched bright light in order to improve fatigue and quality of life.

DETAILED DESCRIPTION:
After a BI , patients complain in particular about sequel fatigue. This symptom affects about 50 % of the patients; it is severe, with a repercussion on quality of life, reeducation and occupational reintegration, and persists often at a distance of the accident. The investigators' hypothesis is that patients who presented a severe BI could benefit from a treatment by blue enriched withe bright light in order to improve fatigue and quality of life.

The main objective is to decrease fatigue and the secondary objectives are to improve quality of life,decrease daytime sleepiness and increase vigilance.

This is a randomized clinical trial with 2 groups blue enriched withe bright light versus nothing) including 20 patients.The treatment will take 8 weeks with 30 minutes exposition at awakening to withe blue enriched bright light (Luminette, Belgium). The investigators willl estimate the fatigue severity scale score , the quality of life the score (SF12), the sleepiness Epworth score, and the Psychomotor Vigilance Task (PVT) The investigators will included patient with severe BI more than six months after the BI.

ELIGIBILITY:
Inclusion Criteria:

* Severe brain injury patients more than 6 months after the trauma
* Out of the phase of post-traumatic amnesia (score in Galveston Orientation and Amnesia Test (GOAT) upper to 75)
* Initial score on the Glasgow coma scale inferior or equal to 8 within the first 24 hours after brain injury, except sedation
* Age from 18 to 65 years old
* Fatigue severity score ( FSS) superior or equal to 4 and/or a score on the sleepiness Epworth scale superior or equal to 10 and/or a score to the quality questionnaire of sleep of Pittsburg > in 5
* Having given a writing informed consent
* Registered on the Social Security

Exclusion Criteria:

* Non-stabilized psychiatric neurological affection and/or endocrine diseases or drug addiction
* Major depression diagnosed with the "MINI" depression scale
* Cognitive, behavioural or motor disorders incompatible with use of phototherapy glasses
* Night workers or transméridien journey in the last month
* Chronic fatigue syndrome before the accident
* Deafness
* Major obesity (BMI > 33)
* High risk of apnea syndrome in the Berlin questionnaire
* Consumption of long half-l hypnotics or stimulants
* Treatments with antidepressants are tolerated if the dose is stable during all the participation on approval and for at least one month before the inclusion.
* Eye lesion, in particular of the retina
* Photosensibility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 30 minutes
  Fatigue measure by fatigue severity scale

SECONDARY OUTCOMES:
Epworth slumber scale | 30 minutes
  Subjective Slumber measured by Epworth slumber scale
Analog visual scales | 10 minutes
  subjective slumber measured by Epworth slumber scale
Psychomotor Vigilance Task | 15 minutes
  vigilance measured by Psychomotor Vigilance Task
P300 | 30 minutes
  Cognitive evoked potential measure by P300

CONTACTS AND LOCATIONS:
Overall Officials: MARIA ANTONIA QUERA SALVA, MD PhD, Principal Investigator — RAYMOND POINCARE HOSPITAL; SARAH HARTLEY, MD, Study Chair — RAYMOND POINCARE HOSPITAL
Locations (1):
- Hopital Raymond Poincare, Garches, France

REFERENCES:
- [Derived] Quera Salva MA, Azabou E, Hartley S, Sauvagnac R, Leotard A, Vaugier I, Pradat Diehl P, Vallat-Azouvi C, Barbot F, Azouvi P. Blue-Enriched White Light Therapy Reduces Fatigue in Survivors of Severe Traumatic Brain Injury: A Randomized Controlled Trial. J Head Trauma Rehabil. 2020 Mar/Apr;35(2):E78-E85. doi: 10.1097/HTR.0000000000000500. PMID 31246878